CLINICAL TRIAL: NCT02956863
Title: The Effect of Osteopathic Manipulative Treatment in Pain and Functionality Individuals With Nonspecific Chronic Neck Pain: Randomized Clinical Trial
Brief Title: The Effect of Osteopathic Treatment in Pain and Functionality Individuals With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Brasileiro de Osteopatia (Other)
Responsible Party: Principal Investigator, Sandro Groisman, PT, DO, MSc, DO Ms, Instituto Brasileiro de Osteopatia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Osteopathic; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercises (Active Comparator): Individuals with neck pain will receive a exercises program. Participants will receive treatments during 4 weeks, 1 treatments per week.
  Interventions: Procedure: Exercises
- Osteopathic manipulative treatment (Experimental): Individuals with neck pain in this group will also receive a exercises program and the participants will receive treatments during 4 weeks, 1 treatments per week associated with Osteopathic Manipulative Treatment (OMT)
  Interventions: Procedure: Osteopathic manipulative treatment

INTERVENTIONS:
Procedure: Osteopathic manipulative treatment — Osteopathic manipulative treatment delivered on pragmatic way.
  Arms: Osteopathic manipulative treatment
Procedure: Exercises — Exercise for stretching and strength for neck muscles
  Arms: Exercises

SUMMARY:
The purpose of this study is to determine whether manipulative osteopathic treatment associated exercises improves pain and function in individuals with chronic non-specific neck pain

DETAILED DESCRIPTION:
The purpose of this study is to determine whether manipulative osteopathic treatment associated exercises improves pain and function in individuals with chronic non-specific neck pain Design: a randomized single blind placebo controlled trial will be conducted trial. Patients (n=40) with non-specific neck pain will be randomized to receive 1) osteopathic manipulative treatment and exercise (n=20) or 2) exercise alone (n=20). Participants will receive 8 treatments during 4 weeks.

Clinical outcomes will be obtained at 1 week, four weeks and 24 weeks after end of treatment.

Methods:

The primary outcome will be pain measured by 11-point numerical pain rating scale.

The secondary outcome will be disability measured by the Neck Disability Index, range of motion measured by Cervical Range of Motion device, Pressure pain threshold measured by electronic algometer.

ELIGIBILITY:
Inclusion Criteria:

Symptoms of chronic neck pain does not specify that persists for more than 3 months

Exclusion Criteria:

individuals who report inflammatory previous surgery, spondylolisthesis, spinal stenosis, herniated disc, radiculopathy, fracture and musculoskeletal degenerative diseases. , Cancer, neurological diseases, pregnancy. They will be excluded participants who received some form of manipulative treatment in the last three months.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 30 days after end treatment
  measured by numeric rating scale

SECONDARY OUTCOMES:
range of motion | 30 days after end treatment
  measured by CROM device
Pressure pain threshold | 30 days after end treatment
  measured by electronic algometer
functionality and disability | 30 days after end treatment
  measured by Neck Disability Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Groisman, MS, Principal Investigator — IBO Brazilian Osteopathic Institute
Locations (1):
- Sandro Groisman, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No